CLINICAL TRIAL: NCT01609816
Title: Phase I Study of Dasatinib in Recipients of Autologous Stem Cell Transplantation for Hematologic Malignancies.
Brief Title: Dasatinib for Modulating Immune System After Autologous Stem Cell Transplants for Multiple Myeloma, Non-Hodgkin, or Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual. No Analyses were performed
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Abhinav Deol, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-203
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Non-Hodgkin's Lymphoma; Multiple; Mycosis Fungoides; Hodgkin's Lymphoma; Multiple Myeloma
Keywords: adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; cutaneous B-cell non-Hodgkin lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; hepatosplenic T-cell lymphoma; intraocular lymphoma; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncutaneous extranodal lymphoma; peripheral T-cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent small lymphocytic lymphoma; refractory hairy cell leukemia; refractory multiple myeloma; small intestine lymphoma; splenic marginal zone lymphoma; stage I adult Burkitt lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult Hodgkin lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult T-cell leukemia/lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I mantle cell lymphoma; stage I marginal zone lymphoma; stage I multiple myeloma; stage I small lymphocytic lymphoma; stage IA mycosis fungoides/Sezary syndrome; stage IB mycosis fungoides/Sezary syndrome; stage II adult Hodgkin lymphoma; stage II adult T-cell leukemia/lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage II multiple myeloma; stage IIA mycosis fungoides/Sezary syndrome; stage IIB mycosis fungoides/Sezary syndrome; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult T-cell leukemia/lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III multiple myeloma; stage III small lymphocytic lymphoma; stage IIIA mycosis fungoides/Sezary syndrome; stage IIIB mycosis fungoides/Sezary syndrome; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult T-cell leukemia/lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IVA mycosis fungoides/Sezary syndrome; stage IVB mycosis fungoides/Sezary syndrome; T-cell large granular lymphocyte leukemia; testicular lymphoma; Waldenström macroglobulinemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Mycosis Fungoides; Hodgkin Disease; Multiple Myeloma; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasatinib (Experimental): This is a phase 1 dose escalation study, using a standard 3+3 design. Dasatinib is administered orally once daily in the outpatient setting. The starting dose of dasatinib is 20 mg daily. The increment of dose escalation is 20 mg per dose level. Thus, there will be 5 dose levels (20 mg, 40 mg, 60 mg, 80 mg and 100 mg, respectively) with 3 patients in each cohort. Patients will continue on dasatinib for 6 months
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Patients receive dasatinib PO every day (QD) for 6 months.
  Other Names: BMS-354825; Sprycel

SUMMARY:
This study uses a drug called dasatinib to produce an anti-cancer effect called large granular lymphocyte cellular expansion. Large granular lymphocytes are blood cells known as natural killer cells that remove cancer cells. Researchers think that dasatinib may cause large granular lymphocyte expansion to happen in patients who have received a blood stem cell transplant (SCT) between 3 to 15 months after the blood SCT. In this research study, researchers want to find how well dasatinib can be tolerated, the best dose to take of dasatinib and to estimate how often large granular lymphocytic cellular expansion happens at the best dose of dasatinib.

DETAILED DESCRIPTION:
This is a phase I, dose-escalation study.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of first ASCT for the treatment of hematologic malignancies (multiple myeloma, Hodgkin's and non Hodgkin's lymphoma)
* Patients must be between 100 to 180 days after ASCT
* Dasatinib use prior to ASCT is allowed
* Performance status >= 60%
* Presence of LGL clone prior to enrollment will not be an exclusion criterion if the LGL clone is < 25% of T cell population
* Total bilirubin < 2.0 times the institutional upper limit of normal (ULN)
* Hepatic enzymes (aspartate aminotransferase [AST], alanine aminotransferase [ALT]) =< 2.5 times the institutional ULN
* Serum creatinine < 1.5 times the institutional ULN
* Hemoglobin >= 8 g/dL
* Absolute neutrophil counts >= 1,500 cells per uL
* Platelets >= 100,000 per uL
* Patient should be able to provide signed written informed consent; before any study procedures are performed, subjects will have the details of the study described to them, and they will be given a written informed consent document to read; then, if subjects consent to participate in the study, they will indicate that consent by signing and dating the informed consent document in the presence of study personnel; written consent will include a Health Insurance Portability and Accountability Act (HIPAA) form according to institutional guidelines
* Patient should be able to take oral medication (dasatinib must be swallowed whole)

Exclusion Criteria:

* Patients who have evidence of disease progression before day 100 after ASCT
* Sex and reproductive status:

  * Women of childbearing potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after the last dose of study drug
  * Women who are pregnant or breastfeeding
  * Women with a positive pregnancy test
  * Sexually active fertile men not using effective birth control if their partners are WOCBP
* Medical history and concurrent diseases:
* No malignancy (other than the one treated in this study) which required radiotherapy or systemic treatment within the past 5 years
* Concurrent medical condition which may increase the risk of toxicity, including:

  * Pleural or pericardial effusion of any grade at the time of screening for study
  * Cardiac symptoms; any of the following should be considered for exclusion:

    * Uncontrolled angina, congestive heart failure or myocardial infarction (MI) (within 6 months)
    * Diagnosed congenital long QT syndrome
    * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
    * Prolonged corrected QT (QTc) interval on pre-entry electrocardiogram (> 450 msec)
* History of significant bleeding disorder unrelated to cancer, including:

  * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)* Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
  * Ongoing or recent (=< 3 months) significant gastrointestinal bleeding
* Any previous history of >= grade 3 toxicity to dasatinib
* Prohibited treatments and or therapies
* Category I drugs that are generally accepted to have a risk of causing torsades de pointes including: (patients must discontinue drug 7 days prior to starting dasatinib):

  * Quinidine, procainamide, disopyramide
  * Amiodarone, sotalol, ibutilide, dofetilide
  * Erythromycin, clarithromycin
  * Chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
  * Cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine
* Patient agrees to discontinue St. Johns Wort while receiving dasatinib therapy (discontinue St. Johns Wort at least 5 days before starting dasatinib)
* Patient agrees that intravenous (IV) bisphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia
* Other exclusion criteria:
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-02-12 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) graded according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version 4 | 2 months
Maximum tolerated dose (MTD)graded according to the NCI CTCAE version 4 | 2 months
  Defined as highest dose at which no more than one of dose limiting toxicity (DLT) is observed (among the first 6 patients treated and evaluable for toxicity for the purpose of cohort dose escalation decisions).

SECONDARY OUTCOMES:
Incidence of large granular lymphocytes (LGL) lymphocytosis | 6 months
  95% confidence intervals estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Abhinav Deol, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT01609816/Prot_SAP_000.pdf